CLINICAL TRIAL: NCT06907953
Title: CZI Rare As One: Co-designing an App and Wearable Based Compass for Rare Diseases
Status: Completed | Type: Observational
Sponsor: 4YouandMe (Other)
Collaborators: Patient Led Research Collaborative (PLRC) (Unknown); Mission: Cure (Other); Cure VCP Disease (Unknown); Foundation for Sarcoidosis Research (FSR) (Unknown); Primary Ciliary Disease Foundation (PCD) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 4UCZIRAO
Record Dates: First submitted 2025-01-31; First posted 2025-04-03 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Pancreatitis, Chronic; Sarcoidosis; VCP Disease; Long COVID; PCD; Symptoms and Signs; Wearables
MeSH Terms: conditions — Pancreatitis, Chronic; Sarcoidosis; Post-Acute COVID-19 Syndrome; Signs and Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Other: Observational - no intervention — Pilot, observational study - no intervention

SUMMARY:
The CZI Rare As One study is a Chan Zuckerberg Initiative funded study that aims to co-design and pilot test unique symptom tracking and transmitting apps across 5 different sub-arms that includes individuals with Long COVID, Pancreatitis, Sarcoidosis, Vasolin-Containing Protein (VCP) disease and Primary Ciliary disease (PCD). This study aims to use multimodal digital health tools to enable patients to self-monitor their symptoms in passive and active ways.

DETAILED DESCRIPTION:
The CZI Rare As One Study is a pilot, beta testing that aims to recruit ~50 participants per disease group (LongCOVID, pancreatitis, sarcoidosis, VCP disease, and PCD) totalling 250 participants. Participants will be instructed to us a co-designed study app alongside specific wearable and smart devices as outlined below for 5 months.

LongCOVID: Oura ring, Empatica EmbracePlus wristband, Lumia ear device Pancreatitis: Oura ring, Empatica EmbracePlus wristband Sarcoidosis: Oura ring VCP Disease: Oura ring, MIR Smart One Spirometer, Apple Watch series 8 PCD: Oura ring, MIR Smart One Spirometer

Research staff (engagement specialists) will check-in via phone every 2 weeks with participants to provide support, troubleshoot tech problems, solicit study-related feedback and collect context related information about the participants disease.

The study app collects symptom specific information for each disease group, measures of disease burden, quality of life, and information about participants routines through self-reported surveys and tasks (cognitive, active tasks) and passive phone metadata derived from SensorKit's Research framework and an Android equivalent framework.

ELIGIBILITY:
GENERAL INCLUSION CRITERIA

* 18+ years (except 14+ years for the PCD sub-arm)
* own a personal mobile device and use this phone to download and use the app for the study
* resides in the US
* be willing to use the study wearable devices
* have a clinician confirmed or suspected diagnosis of one of the 5 rare conditions as defined below in the cohort specific inclusion criteria below:

Long COVID sub-arm:

* have experienced Long COVID for at least 3 months as a continuous, relapsing and remitting, or progressive condition; and
* have experienced within the past week at least one or more of the following symptoms that started or significantly worsened following a COVID infection: shortness of breath, cough, persistent fatigue, post-exertional malaise (worsening of symptoms or fatigue after minimal activity), difficulty concentrating, memory changes, recurring headache, lightheadedness, fast heart rate, sleep disturbance, problems with taste or smell, bloating, constipation, and diarrhea.
* symptom(s) of COVID significantly impact your ability to work, ability to give care, enjoy recreational activities or reduce your quality of life
* Own a personal iPhone 8 (iOS 16+) or Android smartphone (version 12 or newer)

Sarcoidosis sub-arm

* have a diagnosis of sarcoidosis confirmed by a doctor, and have experienced fatigue for at least 2 days in the past month
* Own a personal iPhone 6s (iOS 15+) or Android smartphone (version 12 or newer)

Pancreatitis sub-arm

* have a diagnosis of chronic pancreatitis confirmed by a doctor, have had at least 1 pancreatitis flare in the past year, and have not had a surgery that completely removed the pancreas
* Own a personal iPhone 6s (iOS 15+) or Android smartphone (version 12 or newer)

VCP disease sub-arm

* have a clinician confirmed pathogenic VCP mutation or a family history of VCP disease, and are experiencing symptoms associated with the disease
* Own a personal iPhone 8 (iOS 16+) or Android smartphone (version 12 or newer)

PCD sub-arm

* a genetic test that confirms two abnormal copies (one on each gene) of a gene associated with PCD. These abnormalities must be classified as "pathogenic" or "likely pathogenic."; Or an abnormal electron microscopy cilia biopsy done in a PCD center.; and symptoms consistent with PCD.
* Own a personal iPhone 8 (iOS 16+) or Android smartphone (version 12 or newer)

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a clinician confirmed diagnosis of pancreatitis, sarcoidosis, PCD, VCP disease and LongCOVID (suspected diagnosis).
Sampling Method: Non-Probability Sample
Enrollment: 239 (Actual)
Dates: Start 2025-02-06 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Retention | 5 months
  Proportion of participants retained for the full study
Adherence | 5 months
  Average adherence of daily app use surveys/tasks over follow-up

SECONDARY OUTCOMES:
Usability | 5 months
  Patient reported usability of study devices (qualitative). Participants will be asked over bi-weekly phone check-in calls a number of questions relating to study experience outlined below. Qualitative synthesis of this unstructured text will be completed to understand themes.
  IS THERE ANYTHING THAT IS PARTICULARLY MAKING YOU WANT TO USE THE STUDY APP LESS? IS THERE ANYTHING ABOUT THE STUDY APP THAT YOU DIDN'T EXPECT TO ENJOY BUT YOU DO? WHAT ARE THE PRIMARY BARRIERS TO USING THE STUDY APP? 1 FORGETFULNESS; 2 INCONVENIENCE; 3 HEALTH-RELATED BARRIERS; 4 ENVIRONMENTAL BARRIERS; 5 TECHNOLOGICAL BARRIERS; 6 DIGITAL LITERACY; 7 TASK FATIGUE; 8 LOW PERCEIVED UTILITY; 9 PRIVACY & CONFIDENTIALITY CONCERNS; 10 OTHER
  WHAT ARE THE PRIMARY BARRIERS TO USING THE OURA RING?
  1 FORGETFULNESS; 2 INCONVENIENCE; 3 HEALTH-RELATED BARRIERS; 4 ENVIRONMENTAL BARRIERS; 5 TECHNOLOGICAL BARRIERS; 6 DIGITAL LITERACY; 7 TASK FATIGUE; 8 LOW PERCEIVED UTILITY; 9 PRIVACY & CONFIDENTIALITY CONCERNS; 10 OTHER
Benefits/Harms | 5 months
  Patient reported benefits and harms from using the study devices (qualitative). Participants will be asked over bi-weekly phone check-in calls a number of questions relating to study experience outlined below. Qualitative synthesis of this unstructured text will be completed to understand themes.
  ARE THERE ANY FEATURES OF THE STUDY APP THAT YOU ARE FINDING BENEFICIAL TO YOUR HEALTH / WELLNESS ?
  ARE THERE ANY FEATURES OF THE STUDY APP THAT YOU ARE FINDING NOT BENEFICIAL / HARMFUL TO YOUR HEALTH / WELLNESS ?
  ARE THERE ANY FEATURES OF THE OURA RING / OURA APP THAT YOU ARE FINDING BENEFICIAL TO YOUR HEALTH / WELLNESS ?
  ARE THERE ANY FEATURES OF THE OURA RING / OURA APP THAT YOU ARE FINDING NOT BENEFICIAL / HARMFUL TO YOUR HEALTH / WELLNESS ?

CONTACTS AND LOCATIONS:
Locations (1):
- 4YouandMe, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All data, source code, and study findings will be made open source via public repositories (TBD), GitHub, and published documents.
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: 1 year of study completion
Access Criteria: All qualified researchers with an approved IRB protocol
URL: http://4youandme.org